CLINICAL TRIAL: NCT06679231
Title: Improving Patient Experience in Gynecologic Examinations With a Stress Ball: A Randomized Controlled Trial
Brief Title: Stress Balls in Gynecologic Exams: A Patient Comfort Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betul Uncu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-95531838-050.99-116026
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-11

CONDITIONS: Gynecologic
Keywords: pain; women health; pap-smear; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stress Ball (Experimental): After the initial measurements of the participants assigned to the experimental group, the students involved in the project will accompany the patient and prepare the patient for the gynecological examination. To make the patient feel more comfortable during the gynecological examination, she will be given two stress balls. The patient will be asked to count each time she squeezes the stress ball during the examination. During the gynecological procedure, the participant will be administered the first EC-3. The stress ball intervention will help to reduce the participant's anxiety level and make the examination process more tolerable.
  Interventions: Behavioral: Stress Ball
- Control (No Intervention): After the initial measurements of the participants assigned to the control group, the student involved in the project will prepare the patient for a gynecological examination. Patients in the control group will be provided with only a relaxing environment, without a stress ball during the examination.

INTERVENTIONS:
Behavioral: Stress Ball — After the initial measurements of the participants assigned to the experimental group, the students involved in the project will accompany the patient and prepare the patient for the gynecological examination. To make the patient feel more comfortable during the gynecological examination, she will be given two stress balls. The patient will be asked to count each time she squeezes the stress ball during the examination. During the gynecological procedure, the participant will be administered the first EC-3. The stress ball intervention will help to reduce the participant's anxiety level and make the examination process more tolerable. In addition, the student's support to the patient will make the examination more comfortable and contribute to the participant's psychological well-being.
  Arms: Stress Ball

SUMMARY:
Women's anxiety about gynecological examinations causes them to skip examinations during this process. Research shows that women with high levels of anxiety are more likely to feel pain. Women who can manage their anxiety can increase their satisfaction by reducing pain levels during the examination . The stress ball has the potential to improve the patient experience by reducing these anxieties. This will positively affect women's willingness to participate in gynecological examinations and follow-up processes.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35,
* Being literate, knowing and understanding Turkish,
* Don't have a pap-smear test for the first time,

Exclusion Criteria:

* Presence of chronic pain in the pelvic region,
* Presence of a condition in the wrists that prevents squeezing the stress ball,
* Congenital malformation of the cervix, .Having a known diagnosis of a serious psychiatric illness.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — suitable for women who have had a pap smear
Enrollment: 141 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Reduction of pain | 30 minutes after application
  pain assessed by VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı Training and Research Hospital, Ağrı, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen L, Lamarche L, Lennox R, Ramdyal A, Patel T, Black M, Mangin D. Strategies to Mitigate Anxiety and Pain in Intrauterine Device Insertion: A Systematic Review. J Obstet Gynaecol Can. 2020 Sep;42(9):1138-1146.e2. doi: 10.1016/j.jogc.2019.09.014. Epub 2019 Dec 25. PMID 31882291